CLINICAL TRIAL: NCT04718272
Title: Safety and Feasibility of the Application of Thoracic Puncture Tube VS Combination of Puncture Tube and Silicone Tube After Uniportal VATS Pulmonary Lobectomy
Brief Title: Safety and Feasibility of the Application of Thoracic Puncture Tube After Pulmonary Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDTM UNION
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Chest Tubes; Pneumonectomy; Minimally Invasive Surgery
Keywords: Chest Tubes; Pneumonectomy; Minimally Invasive Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puncture tube group (Experimental): After the operation, the traditional traditional silicone tube which placed through the surgical incision was removed in the operating room, and the small puncture tube was retained for thoracic drainage.
  Interventions: Procedure: thoracic drainage management
- Traditional tubes group (No Intervention): Routine thoracic drainage management measures were adopted, that is, both of the small puncture tube and traditional silicone tube were retained after surgery.

INTERVENTIONS:
Procedure: thoracic drainage management — After uniportal VATS pulmonary lobectomy, the traditional silicone tube which placed through the surgical incision was removed in the operating room in the experimental group.
  Arms: Puncture tube group

SUMMARY:
There have been several reports on the feasibility of a no-drain policy after pneumonectomy, but the policy is not widely accepted because silent massive hemorrhage, delayed air leaks, and chylothorax would always be major worries for thoracic surgeons, and all of the researches were retrospective case studies with small sample size and insufficient evidence. Therefore, the purpose of this study is to to evaluate safety and feasibility of an improved policy, the application of a small thoracic puncture tube after pulmonary lobectomy.

DETAILED DESCRIPTION:
This study will be accepted in patients with uniportal VATS(Video-assisted Thoracoscopic Surgery）lobetomy. A randomized controlled study protocol will be used, and The patients will be devided into two groups: experimental group for the application of a small thoracic puncture tube and control group for the application of Combination of the puncture tube and traditional silicone tube. The intraoperative conditions, postoperative recovery and the incidence of perioperative complications will be compared. The safety and feasibility of the application of the small thoracic puncture tube after pulmonary lobectomy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18-70 years old, male and female unlimited;
2. Cardiopulmonary function can tolerate operation;
3. Primary non-small cell lung cancer was diagnosed by preoperative or intraoperative pathology. The surgical ranges are uni-portal VATS lobectomy with or without mediastinal lymph node dissection or sampling. In cases with multiple nodules in other lobes of the same side, small wedge resections are allowed;
4. No air leakage was observed intraoperatively. Meanwhile, after operation, there are also no air leakage observed in water seal bottle when patients are changed from lateral decubitus to horizontal position.
5. Patients and their family members can understand and are willing to participate in this clinical study and sign the informed consent..

Exclusion Criteria:

1. Patients with a severe emphysema or pulmonary bullae;
2. Patients with a history of chemotherapy or chemo-radiotherapy;
3. Patients with a history of chest surgery;
4. Extensive thoracic adhesion ;
5. A history of serious mental illness;
6. Patients with other conditions considered by the researcher should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complications | within 30 days after surgery
  The incidence of complications within 30 days after surgery in each arm

SECONDARY OUTCOMES:
Incidence of subcutaneous emphysema after operation | within 30 days after surgery
  The incidence of subcutaneous emphysema after operation in each arm
Incidence of postoperative pneumothorax | within 30 days after surgery
  The incidence of postoperative pneumothorax in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chen, MD, Study Director — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China